CLINICAL TRIAL: NCT02743832
Title: A Randomized，Multicenter，Prospectie，Controlled Clinical Study on Tumor Budding Guiding Individualized Surgical Planning of Early-stage Oral Squamous Cell Carcinoma.
Brief Title: A Study on Tumor Budding Guiding Individualized Surgical Planning of Early-stage Oral Squamous Cell Carcinoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinsong Hou (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); Hospital of Stomatology, Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Jinsong Hou, Vice Director, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HouJ-2015018
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Oral squamous cell carcinoma; Tumor budding; Cervical lymph node dissection
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-level tumor budding group with CLND (Experimental): Resection for primary lesion and cervical lymph node dissection (CLND) are performed in the early-stage oral squamous cell carcinoma which tumor budding is a high level.
  Interventions: Procedure: Resection for primary lesion and cervical lymph node dissection
- High-level tumor budding group without CLND (Experimental): Only resection for primary lesion is performed in the early-stage oral squamous cell carcinoma which tumor budding is a high level.
  Interventions: Procedure: Resection for primary lesion only
- Low-level tumor budding group with CLND (Experimental): Resection for primary lesion and cervical lymph node dissection (CLND) are performed in the early-stage oral squamous cell carcinoma which tumor budding is a low level.
  Interventions: Procedure: Resection for primary lesion and cervical lymph node dissection
- Low-level tumor budding group without CLND (Experimental): Only resection for primary lesion is performed in the early-stage oral squamous cell carcinoma which tumor budding is a low level.
  Interventions: Procedure: Resection for primary lesion only

INTERVENTIONS:
Procedure: Resection for primary lesion and cervical lymph node dissection — Resection for primary lesion and cervical lymph node dissection are performed in the early-stage oral squamous cell carcinoma.
  Arms: High-level tumor budding group with CLND; Low-level tumor budding group with CLND
Procedure: Resection for primary lesion only — Only resection for primary lesion is performed in the early-stage oral squamous cell carcinoma.
  Arms: High-level tumor budding group without CLND; Low-level tumor budding group without CLND

SUMMARY:
The purpose of this study is to determine whether cervical lymph node dissection is necessarily performed in the presence of early-stage oral squamous cell carcinoma.

DETAILED DESCRIPTION:
Oral squamous cell carcinoma is the most common malignant tumor of oral and maxillofacial region, and prone to early cervical lymph node metastases. Lymphatic spread is associated with increased risk of loco-regional recurrence, therefore, the identification of lymph node metastases preoperatively is very important for the optimal surgical therapy. Recently, cervical lymph node dissection(CLND) is performed in the presence of oral squamous cell carcinoma. However, whether cervical lymph node dissection is necessarily performed in the presence of early-stage oral squamous cell carcinoma is still controversial. CLND will represent over-treatment in some case of early-stage oral squamous cell carcinoma. Therefore, How to accurately predict whether a patient should be performed CLND is important. Our previous study show that tumor budding is closely related to lymphatic spread in the oral squamous cell carcinoma. The purpose of this study is to find that whether the tumor budding guide the individualized surgical planning of early-stage oral squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Han race;
2. Oral squamous cell carcinoma is confirmed by pathology;
3. The section of oral squamous cell carcinoma including primary two-thirds prior to the tongue, buccal mucosa， gingiva， mouth floor， hard palate mucosa;
4. The primary lesion is no more than 4cm;
5. Do not find cervical lymph node metastases and distant metastasis in the clinical examination including physical examination and MRI;
6. Patients and families agree to participate in the study;
7. Patients do not have cognitive disorders.

Exclusion Criteria:

1. Do not meet the inclusion criteria;
2. The primary lesion is more than 4cm or invade adjacent tissues;
3. Do not review on schedule;
4. Patients receive not only surgical procedures, but other antineoplastic treatment;
5. There are serious adverse events after operation;
6. Patients quit the study voluntarily;
7. Patients quit the study because of physical condition.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2022-09-04 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Five-year survival rate | After the first year, review every three months at a time；The next four years, review every six months at a time.
  The time from the first operation to death was recorded
Disease free survival | After the first year, review every three months at a time；The next four years, review every six months at a time.
  The time from the start of surgery to the discovery of the first cervical lymphatic metastases

SECONDARY OUTCOMES:
Recurrence rate | After the first year, review every three months at a time；The next four years, review every six months at a time.
  To investigate the local recurrence rate and the recurrence rate of cervical lymphatic metastasis.
Evaluation of quality of life | After the first year, review every three months at a time；The next four years, review every six months at a time.
  Complete the University of Washington Quality of Life Form (UW-QOL) To understand the quality of life of patients after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Hou, PhD, Study Director — Guanghua School of Stomatology, Hospital of Stomatolagy Sun Yat-sen University
Locations (1):
- Guanghua School of Stomatolagy, Hospital of Stomatology Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Almangush A, Salo T, Hagstrom J, Leivo I. Tumour budding in head and neck squamous cell carcinoma - a systematic review. Histopathology. 2014 Nov;65(5):587-94. doi: 10.1111/his.12471. Epub 2014 Oct 6. PMID 24897954
- [Result] Almangush A, Bello IO, Keski-Santti H, Makinen LK, Kauppila JH, Pukkila M, Hagstrom J, Laranne J, Tommola S, Nieminen O, Soini Y, Kosma VM, Koivunen P, Grenman R, Leivo I, Salo T. Depth of invasion, tumor budding, and worst pattern of invasion: prognostic indicators in early-stage oral tongue cancer. Head Neck. 2014 Jun;36(6):811-8. doi: 10.1002/hed.23380. Epub 2013 Sep 2. PMID 23696499
- [Result] Da Sacco L, Masotti A. Recent insights and novel bioinformatics tools to understand the role of microRNAs binding to 5' untranslated region. Int J Mol Sci. 2012 Dec 27;14(1):480-95. doi: 10.3390/ijms14010480. PMID 23271365
- [Result] Xie N, Wang C, Liu X, Li R, Hou J, Chen X, Huang H. Tumor budding correlates with occult cervical lymph node metastasis and poor prognosis in clinical early-stage tongue squamous cell carcinoma. J Oral Pathol Med. 2015 Apr;44(4):266-72. doi: 10.1111/jop.12242. Epub 2014 Aug 28. PMID 25169851
- [Result] Hori Y, Kubota A, Yokose T, Furukawa M, Matsushita T, Takita M, Mitsunaga S, Mizoguchi N, Nonaka T, Nakayama Y, Oridate N. Predictive Significance of Tumor Depth and Budding for Late Lymph Node Metastases in Patients with Clinical N0 Early Oral Tongue Carcinoma. Head Neck Pathol. 2017 Dec;11(4):477-486. doi: 10.1007/s12105-017-0814-1. Epub 2017 Apr 3. PMID 28374102